CLINICAL TRIAL: NCT04198610
Title: Evaluation and Correlation of Serum Fetuin-A Levels in Periodontal Health and Disease: A Clinico-biochemical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_63396
Record Dates: First submitted 2019-02-26; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-02

CONDITIONS: Gingivitis and Periodontal Diseases
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy (No Intervention): Ten patients with clinically healthy gingiva with probing depth less than 3mm and less than or equal to 10% sites with gingival bleeding on probing present.
- chronic gingivitis (No Intervention): Chronic gingivitis was defined as having probing depth (PD) less than or equal to 4mm, relative attachment loss (RAL) ) less than or equal to 3mm and more than to 25% sites with gingival bleeding present (BOP)
- chronic periodontitis (Active Comparator): Chronic periodontitis was defined as having probing depth more than or equal to 5mm, RAL more than or equal to 8mm, with more than or equal to 10% sites with BOP positive and evidence of bone loss determined radiographically.
  Non surgical periodontal therapy (SRP) was concluded in 3 months. Within the duration of the study, all subjects received supportive therapy
  Interventions: Procedure: Non surgical periodontal therapy

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — Procedure/Surgery: non surgical periodontal therapy and root planing (SRP) was performed in two to four appointments lasting approximately 60 minutes each under local anaesthesia (2% lignocaine hydrochloride with 1:2,00,000 adrenaline) using area specific Gracey periodontal curettes and an ultrasonic device. The treatment was concluded in 3 months. Within the duration of the study, all subjects received supportive therapy, which included professional plaque control and reinstruction of oral hygiene.
  Arms: chronic periodontitis

SUMMARY:
The present clinico-biochemical study was carried out to estimate the levels of Fetuin A and MMP7 in serum of systemically healthy subjects in periodontal health and disease and to evaluate the impact of periodontal interventional therapy (scaling and root planing) on the same.

DETAILED DESCRIPTION:
Sixty sex-matched subjects (30 males and 30 females) belonging to a common age group (30-39 yrs) were enrolled for the study to eliminate bias from confounding factors. They were divided into three groups consisting of 20 subjects in each group based on the clinical and radiological parameters; Periodontally healthy (Group I), Chronic gingivitis (Group II) and chronic periodontitis ( Group IIIa) from whom serum samples were collected. The Group IIIb further comprised of the subjects from Group IIIa, who had received non-surgical periodontal therapy (scaling and root planing). Serum samples were collected at baseline and at 12 weeks post therapy. Fetuin A and MMP-7 concentration was determined from serum samples of patients using ELISA. The results of our study depicted that Fetuin A concentration negatively correlates, whereas, MMP7 positively correlates with the extent of periodontal inflammation. Further, Periodontal therapy demonstrated a significant increase in serum Fetuin A and decrease in MMP 7 levels establishing the influence of periodontal therapy in stabilizing their levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age group of 30-39 years.
2. Systemically healthy subjects.
3. Patient who are co-operative and able to attend follow up.
4. Patient who have not received any periodontal treatment within the past six months of baseline examination.
5. Dentition with at least 20 functional teeth.

Exclusion Criteria:

1. Medically compromised patients (history of diabetes mellitus, liver diseases, cardiovascular disease, kidney diseases, rheumatoid arthritis, bone diseases pulmonary disease, viral and fungal infections).
2. Patients with calcification disorders (chronic kidney disease with vascular calcification, hyperparathyroidism, excessive intake of vitamin D, valvular calcific aortic stenosis
3. Aggressive periodontitis.
4. Bleeding disorders
5. Gross oral pathology and suppuration
6. Patients who had received antibiotic therapy and anti inflammatory within the last six months.
7. Anomalies of the immune system.
8. Pregnancy and lactation.

Ages: 30 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
estimate the change in levels of Fetuin A and MMP7 in serum at baseline and 3 months post SRP | Serum collection at baseline and 3 months
  Serum was collected at baseline and 3 months and subjected to ELISA

SECONDARY OUTCOMES:
Modified Gingival index (GI) | At baseline and 3 months
  The index was recorded at only baseline for healthy and gingivitis groups and at baseline and 3 months post therapy for periodontitis group
Relative Attachment level (RAL) | At baseline and 3 months
  The index was recorded at only baseline for healthy and gingivitis groups and at baseline and 3 months post therapy for periodontitis group
Probing Depth (PD) | At baseline and 3 months
  The index was recorded at only baseline for healthy and gingivitis groups and at baseline and 3 months post therapy for periodontitis group
Bleeding on Probing (BOP%) | At baseline and 3 months
  The index was recorded at only baseline for healthy and gingivitis groups and at baseline and 3 months post therapy for periodontitis group
Plaque index (PI) | At baseline and 3 months
  The index was recorded at only baseline for healthy and gingivitis groups and at baseline and 3 months post therapy for periodontitis group

CONTACTS AND LOCATIONS:
Overall Officials: BV Karthikeyan, MDS, Study Director — Krishnadevaraya college of Dental sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided